CLINICAL TRIAL: NCT04582175
Title: A Retrospective, One Center Comparison of Outcomes Between Complete Revascularization by PCI at the Time of PPCI or During the Index Hospital Admission in One Hundred MVD Patients With ST-elevation MI Uncomplicated by Cardiogenic Shock
Brief Title: Comparison Between Two Revascularization Strategies in MVD Patients With Uncomplicated ST-elevation MI
Acronym: Promise
Status: Completed | Type: Observational
Sponsor: University of Oradea (Other)
Responsible Party: Principal Investigator, Nichita-Brendea Mihnea-Traian, MD, University of Oradea
Other Study IDs: Uoradea
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: STEMI
Keywords: PPCI, multivessel coronary artery disease, STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: patients who received complete revascularization by angioplasty during the PPCI
  Interventions: Procedure: angioplasty
- Group B: patients who underwent complete revascularization by angioplasty in a staged procedure
  Interventions: Procedure: angioplasty

INTERVENTIONS:
Procedure: angioplasty — angioplasty of all non-culprit lesions

SUMMARY:
The study aimed to compare major adverse cardiac and cerebrovascular events(MACCE) and mortality at one year between two strategies: complete revascularization including non-culprit lesions percutaneous coronary intervention(PCI) during primary PCI(PPCI) versus complete revascularisation during the same hospital admission in multi-vascular coronary artery disease(MVD) patients presenting with ST-elevation myocardial infarction(STEMI) uncomplicated by cardiogenic shock.

DETAILED DESCRIPTION:
Complete revascularisation in MVD patients with STEMI uncomplicated by cardiogenic shock has been shown to improve outcomes, however the optimal timing of treatment of the non-culprit lesions is not known. The 2018 ESC/EACTS Guidelines on myocardial revascularization states that "routine revascularization of non-IRA (infarct related artery) lesions should be considered in patients with multivessel disease before hospital discharge". Our trial showed that among the fore mentioned patients there was no difference regarding outcomes when using a strategy of complete revascularization with non-culprit lesions PCI during PPCI or during the same hospital admission.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with successful PCI (preferably using a drug-eluting stent) to the culprit lesion for STEMI ( PCI for STEMI should be primary PCI in the first 12 hours after symptom onset) and complete revascularization of non-culprit lesions during the index PPCI procedure or during a different procedure performed before index hospital discharge.
2. Multi-vessel disease defined as at least 1 additional non-infarct related coronary artery lesion that is at least 2.5 mm in diameter that has not been stented as part of the primary PCI and that is amenable to successful treatment with PCI and has:

   * At least 75% diameter stenosis (visual estimation) or
   * At least 50% diameter stenosis (visual estimation) with fractional flow reserve (FFR) ≤ 0.80
3. Age between 18 and 90 years
4. Written informed consent could be obtained from all the patients

Exclusion Criteria:

1. Rescue PCI for failed fibrinolysis or a combination strategy where PCI is performed routinely 3-12 hours after fibrinolysis
2. Cardiogenic shock
3. Non-cardiovascular known co-morbidity reducing life expectancy to < 2 years
4. Any factor precluding 1year follow-up
5. Prior Coronary Artery Bypass Graft (CABG) Surgery
6. A different operator from the previously designated
7. Unable to provide consent for any other reason

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: multivessel patients with STEMI uncomplicated by cardiogenic shock
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
one year all-cause mortality | one year
  death at one year
MACCE at one year | one year
  major adverse cardiac and cerebrovascular events including cardiac death, stroke, symptom-driven revascularization, myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Mihnea-Traian T Nichita-Brendea, MD, Principal Investigator — Spitalul Clinic Judetean de Urgenta Oradea
Locations (1):
- Spitalul Clinic Judetean de Urgenta Oradea, Oradea, Bihor County, Romania

IPD SHARING:
Plan to Share IPD: No